CLINICAL TRIAL: NCT03434275
Title: A Phase 3b, Randomized, Double-Blind, Placebo-Control, Multicenter, Evaluation of the Safety and Efficacy of N1539 Administered Preoperatively in Open Unilateral Total Knee Arthroplasty
Brief Title: Evaluation of Preoperative N1539 in Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-17-025
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative
Keywords: Total Knee Arthroplasty; Pain; Analgesia; N1539; Phase 3b; Knee Replacement
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N1539 30 mg (Experimental): N1539 (meloxicam injection for IV use) 30 mg every 24 hours
  Interventions: Drug: N1539
- IV Placebo (Placebo Comparator): IV Placebo every 24 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N1539 — Once Daily
  Other Names: Intravenous meloxicam
  Arms: N1539 30 mg
Drug: Placebo — Once Daily
  Other Names: Intravenous placebo
  Arms: IV Placebo

SUMMARY:
The primary objective of this study is to assess the effect of preoperative administration of N1539 on opioid consumption in subjects undergoing open unilateral total knee arthroplasty compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Be planned to undergo an elective, primary (no repeat arthroplasties) open unilateral total knee arthroplasty (TKA), and be expected to require IV analgesia, remain in an inpatient setting for ≥24 hours, and receive at least two doses of study drug.
* ASA physical status category 1, 2, or 3.
* Female subjects not pregnant or planning/attempting to become pregnant, not lactating; or commits to the use of an acceptable form of birth control for the duration of the study.
* Have a body mass index <40 kg/m^2

Exclusion Criteria:

* Have a known allergy or hypersensitivity to any study treatment.
* Have a history of previous TKA.
* Has plans for a concurrent surgical procedure (eg, bilateral TKA).
* Has TKA planned to be performed under general anesthesia.
* Have a history of myocardial infarction within the preceding 12 months.
* Have, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant condition that would preclude participation.
* Have active or recent (within 6 months) gastrointestinal ulceration or bleeding.
* Have a known bleeding disorder which may be worsened with the administration of an NSAID.
* Be currently receiving treatment with oral meloxicam (Mobic®) or another NSAID within 48 hours prior to surgery.
* Have previously received N1539/IV meloxicam or received any investigational product within 30 days before dosing with study medication.
* Have undergone or be expected to undergo radiation therapy, chemotherapy, or other biological therapy for cancer treatment, within 60 days prior to screening through last follow-up.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Center, Florence, Alabama
  - Research Center, Mobile, Alabama
  - Research Center, Sheffield, Alabama
  - Research Center, Tempe, Arizona
  - Research Center, Tamarac, Florida
  - Research Center, Vero Beach, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berkowitz RD, Steinfeld R, Sah AP, Mack RJ, McCallum SW, Du W, Black LK, Freyer A, Coyle E. Safety and Efficacy of Perioperative Intravenous Meloxicam for Moderate-to-Severe Pain Management in Total Knee Arthroplasty: A Randomized Clinical Trial. Pain Med. 2021 Jun 4;22(6):1261-1271. doi: 10.1093/pm/pnab016. PMID 33502533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N1539 30 mg | IV Placebo
Started | 98 | 96
Treated | 93 | 88
Completed | 93 | 88
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Population: Safety Population - Subjects who received at least 1 study dose
Groups:
- Total: Total of all reporting groups
Arm/Group | N1539 30 mg | IV Placebo | Total
Number analyzed (Participants) | 93 | 88 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.23) | 65.5 (8.11) | 66.2 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 105
  Male | 39 | 37 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 84 | 79 | 163
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 17 | 35
  White | 74 | 70 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 93 | 88 | 181

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use Hour 0-24
Description: Total use of opioid analgesia, in IV morphine equivalent dose, from Hour 0 through 24.
Time Frame: Up to 24 Hours
Measure: Least Squares Mean (Standard Error); unit: mg morphine equivalent
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 93 | 88
mg morphine equivalent | 18.94 (1.320) | 27.73 (1.371)

ADVERSE EVENTS:
Time Frame: Through 30 days post dose
Arm/Group | N1539 30 mg | IV Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/88
Serious Adverse Events (participants affected / at risk) | 3/93 | 9/88
Other Adverse Events (participants affected / at risk) | 65/93 | 81/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=93) | IV Placebo (N=88)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=93) | IV Placebo (N=88)
Nausea (Gastrointestinal disorders) | 37 (42) | 52 (55)
Vomiting (Gastrointestinal disorders) | 15 (16) | 19 (19)
Hypotension (Cardiac disorders) | 13 (14) | 13 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 10 (10)
Constipation (Gastrointestinal disorders) | 10 (10) | 11 (11)
Dizziness (Nervous system disorders) | 6 (8) | 5 (5)
Pyrexia (Investigations) | 7 (7) | 5 (5)
Hypokalemia (Investigations) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03434275/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03434275/SAP_001.pdf